CLINICAL TRIAL: NCT04976465
Title: Treatment and Clinical Outcomes Among SLE Patients in Pregnancy: A Real World Study
Brief Title: Treatment and Clinical Outcomes Among SLE Patients in Pregnancy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Qiang Shu, Chief Physician, Qilu Hospital of Shandong University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SLE with Pregnancy QiluH
Record Dates: First submitted 2021-06-09; First posted 2021-07-26 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Systemic Lupus Erythematosus; Pregnancy Related
Keywords: Systemic Lupus Erythematosus; Pregnancy Related; clinical features; Risk factors
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined with aPL(+) (Experimental): the antiphospholipid antibodies appear in blood at least once
  Interventions: Drug: Anticoagulation; Drug: Without Anticoagulation
- combined with aPL(-) (Experimental): the antiphospholipid antibodies never appear in blood
  Interventions: Drug: Anticoagulation; Drug: Without Anticoagulation

INTERVENTIONS:
Drug: Anticoagulation — Drug:
  1. Prednisone 5-30mg, po, once per day(Qd) prescribed if needed and adjusted due to patient response Other Names: Pred
  2. Hydroxychloroquine 100-200mg, po, twice per day (Bid) prescribed if needed and adjusted due to patient response.
     Other Names: HCQ
  3. Aspirin 100mg, po, once per day (Qd) prescribed if needed and adjusted due to patient response to 32 weeks of pregnancy. 75mg po, once per day (Qd) to 34 weeks of pregnancy. 50mg po, once per day (Qd) to 36 weeks of pregnancy.
     Other Names: Asp
  4. Low molecular weight heparin Enoxaparin 40-60mg, ih, Subcutaneous injection, once per day (Qd) or twice per day (Bid) if needed and adjusted due to patient response.
  Other Names: LMWH
Drug: Without Anticoagulation — Drug:
  1. Prednisone 5-30mg, po, once per day(Qd) prescribed if needed and adjusted due to patient response Other Names: Pred
  2. Hydroxychloroquine 100-200mg, po, twice per day (Bid) prescribed if needed and adjusted due to patient response.
  Other Names: HCQ

SUMMARY:
Systemic lupus erythematosus (SLE) is a kind of systemic autoimmune disease which can cause multiple organs and system damage, which often occurs in women of childbearing age. Compared with healthy pregnant women, SLE patients have higher incidence of premature delivery, preeclampsia and fetal loss during pregnancy. Since SLE patients usually have disease activity during pregnancy and postpartum, and a variety of maternal and fetal diseases are closely related to SLE, it is very important to monitor the disease activity and drug treatment of SLE patients during pregnancy.

DETAILED DESCRIPTION:
Objective: To study the risk factors of poor pregnancy outcomes in SLE patients, and evaluate impact of different therapies on the maternal and fetal health. Methods: Our department and Shanghai Gothic Network Technology Co., Ltd. jointly established the chronic disease management of SLE patients during pregnancy and lactation by using Smart System of Disease Management#SSDM#. With this platform#patients in pregnancy can consult with rheumatologists face to face and follow-up regularly.

Follow-up: Consultation and followup will be scheduled every 4 weeks from confirmed pregnancy until delivery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with systemic lupus erythematosus (SLE) (ACR criteria, 1997);
2. Pregnant women aged 20-45 years old;
3. Willing to participate in this study, willing to medication and follow-up according to the treatment plan, and sign the informed consent.

Exclusion Criteria:

1. The cause of previous abortion was known:

   * Known chromosomal abnormalities in the parent, maternal or embryo.

     - Page 3 of 4 [DRAFT] -• Endocrine dysfunction of pregnant women: luteal dysfunction; Polycystic ovarian syndrome; Ovarian premature failure (FSH

     ≥ 20uu/ L) in follicular stage;
   * Hyperprolactinemia thyroid disease; Other hypothalamic pituitary adrenal axis abnormalities in diabetes mellitus.
   * Abnormal anatomy of pregnant women: abnormal uterus; Asherman syndrome; The uterine fibrosis of cervical insufficiency is more than 5 cm. Vaginal infection.
   * Any known serious heart disease, liver, kidney, blood or endocrine disease.
2. Any active infection Active viral hepatitis includes hepatitis B virus (HBV), hepatitis C virus (HCV), human papillomavirus (HPV). Active infections include small intestine herpes zoster virus (VZV), human immunodeficiency virus (HIV), syphilis or tuberculosis.
3. Allergic to prednisone, hydroxychloroquine, low molecular weight heparin or aspirin.
4. The history of the disease is as follows:

   * There was a history of peptic ulcer or upper gastrointestinal bleeding in the past.
   * The past history of malignant tumor.
   * The past history of epilepsy or psychosis.
5. Women who disagree or cannot complete the follow-up during pregnancy and after delivery.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Live birth rate | After 28 weeks of gestation]
  Percentage of all patients that lead to live birth after 28 weeks of gestation

SECONDARY OUTCOMES:
Early miscarriage | within 10 weeks of gestation]
  Spontaneous pregnancy loss within 10 weeks of gestation
Intrauterine deaths | after 10 weeks of gestation
  Spontaneous pregnancy loss after 10 weeks of gestation
Stillbirth | after 20 weeks of gestation
  Spontaneous pregnancy loss after 20 weeks of gestation
Intrauterine growth retardation (IUGR) | between 28 and 37 weeks of gestation
  weight below the 10th percentile for the gestational age
Number of participants with low amniotic fluid during pregnancy | during pregnancy#an average of 10 months
  the number of participants whose B-ultrasound indicates low amniotic fluid during pregnancy
Number of participants with abnormal S / D values during pregnancy | during pregnancy#an average of 10 months
  the number of participants whose B-ultrasound indicates abnormal S / D values during pregnancy

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoyun Yang, Dr., Study Director — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital, Jinan, Shandong, China